CLINICAL TRIAL: NCT06642727
Title: The Effect of Laughter Yoga on Nurses' Burnout Level and Stress: Randomized Controlled Study
Brief Title: The Effect of Laughter Yoga on Nurses' Burnout Level and Stress
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Ayşe Karataş, student, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-66779070-050.04-2400226440
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Burnout; Stress
Keywords: BURNOUT; stress; nurse; Laughter Yoga
MeSH Terms: conditions — Burnout, Psychological | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: There will be two groups: an experimental group and a control group. The experimental group will undergo laughter yoga, while the control group will not receive any intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the group undergoing laughter yoga (Experimental): Laughter Yoga is a complementary therapy that combines fake and genuine laughter with yoga and breathing exercises, including neck and shoulder exercises. It does not involve humor and is non-pharmacological and non-invasive.
  A session of laughter yoga lasts about 40 minutes and consists of four sections. The first section includes deep breathing exercises, the second section consists of warm-up exercises, the third section involves childlike games, and the fourth section includes laughter exercises.
  The experimental group will consist of 25 participants. Before starting laughter yoga, the "Maslach Burnout Inventory" and the "Nurse Job Stress Scale" will be used to measure burnout and stress levels. Subsequently, a total of eight laughter yoga sessions will be conducted twice a week for one month, after which burnout and stress levels will be measured again using the scales.
  Interventions: Behavioral: laughter yoga
- control group (No Intervention): The control group will consist of 25 participants, whose burnout and stress levels will be measured only using the "Maslach Burnout Inventory" and the "Nurse Job Stress Scale." No intervention will be applied to the participants.

INTERVENTIONS:
Behavioral: laughter yoga — Laughter yoga reduces stress levels through sessions lasting approximately 40 minutes without any invasive or pharmacological interventions. It regulates breathing, relaxes muscles, stimulates circulation, increases pain thresholds, strengthens immunity, lightens the mind, enhances social relationships, promotes mental balance, and boosts self-esteem, hope, energy, and quality of life. The content of a session includes deep breathing exercises, warm-up exercises, childlike games, and laughter exercises.
  Arms: the group undergoing laughter yoga

SUMMARY:
The purpose of this clinical trial is to determine the effect of laughter yoga on the burnout levels and stress of nurses. The main questions of the study are as follows:

1. What is the burnout level of nurses in the control and intervention groups?
2. What is the stress level of nurses in the control and intervention groups?
3. Has there been a change in the burnout levels of nurses practicing laughter yoga?
4. Has there been a change in the stress levels of nurses practicing laughter yoga? To compare whether laughter yoga affects burnout and stress levels, participants will be divided into control and experimental groups. The experimental group will undergo laughter yoga sessions twice a week for one month.

DETAILED DESCRIPTION:
The study examines the stress and burnout levels of nurses and their causes. Stress in nurses arises from factors such as working conditions, compatibility with colleagues, and insufficient equipment, among others. When this stress becomes chronic, it is referred to as burnout. The Maslach Burnout Inventory will be used to assess burnout levels, while the Nurse Stress Scale will be used to assess stress levels. Laughter yoga will be employed as a coping method.

Laughter serves the function of engaging and relaxing effective muscles, improves respiratory functions, regulates blood circulation, reduces stress hormones, boosts the immune system's defenses, raises pain thresholds and tolerance, and enhances mental function. Many studies have observed that the positive effects of laughter yoga on human psychology are beneficial for burnout syndrome. This research will investigate how laughter yoga affects burnout and stress levels.

ELIGIBILITY:
Inclusion Criteria:

* Being a nurse working day and night shifts
* Not having participated in laughter yoga sessions before
* Being willing to participate in the study

Exclusion Criteria:

* Having a physical condition that prevents participation in laughter yoga sessions (hernia, hemorrhoids, vertigo, respiratory disorders, urinary incontinence, epilepsy)
* Not being a nurse
* Working continuously day or continuously night shifts

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Maslach burnout ineventory | 1 month
  The scale consists of 22 items in a 5-point Likert format (0: Never, 1: Very Rarely, 2: Sometimes, 3: Often, 4: Always). It has three dimensions: Emotional Exhaustion (EE, 9 items), Depersonalization (D, 5 items), and Personal Accomplishment Deficiency (PAD, 8 items). EE refers to the emotional overload an individual feels due to their work and is the most significant predictor of burnout. D represents attitudes and behaviors exhibited by the individual without regard to the fact that the people they serve are unique individuals, displaying a lack of emotion. PAD is defined as the inability to cope with problems successfully and feeling insufficient.
  Individuals experiencing burnout are expected to have high scores in EE (0-36), D (0-20), and PAD (0-32). The Cronbach Alpha coefficients for the three subdimensions of the scale are 0.83 for emotional exhaustion, 0.65 for depersonalization, and 0.72 for personal accomplishment deficiency.
Nurse Stress Scale | 1 month
  The original "Nurse Job Stress Scale," developed by Gray-Toft and Anderson, consists of 34 items and seven factors. These factors include: Uncertainty Related to Treatment (8 items = 1,2,3,4,5,6,7,8), Workload (6 items = 9,10,11,12,13,14), Patient Death (5 items = 15,16,17,18,19), Conflict with Physicians (5 items = 20,21,22,23,24), Conflict with Other Nurses (5 items = 25,26,27,28,29), Inadequate Support (3 items = 30,31,32), and Suffering Patient (2 items = 33,34). It is rated using a 4-point Likert system, where (1 point) means never, (2 points) sometimes, (3 points) often, and (4 points) very often. The Cronbach α reliability coefficient of the original scale has been found to be between α = .89 and α = .65 for the subfactors. A high total score indicates that the nurse experiences more frequent periods of stress related to individual stress issues in the physical, psychological, and environmental contexts.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Mustafakemalpaşa Public Hospital, Bursa, Mustafakemalpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No